CLINICAL TRIAL: NCT05115409
Title: Anti-PD-1 Antibody Plus Chidamide and Rituximab Regimen for the Relapsed or Refractory Diffuse Large B Cell Lymphoma (PCR): a Prospective, Multicenter, Single-Arm, Phase II Trial
Brief Title: Anti-PD-1 Antibody Plus Chidamide and Rituximab Regimen in Relapsed or Refractory DLBCL (PCR)
Acronym: PCR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RR-DLBCL-PCR
Record Dates: First submitted 2021-11-09; First posted 2021-11-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Relapsed or Refractory DLBCL
Keywords: DLBCL; Rituximab; Chidamide; Anti-PD-1 Antibody
MeSH Terms: conditions — Recurrence | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 Antibody Plus Chidamide and Rituximab Regimen in Relapsed or Refractory DLBCL (Experimental): Anti-PD-1 Antibody Plus Chidamide and Rituximab Regimen in Relapsed or Refractory DLBCL
  Interventions: Drug: Anti-PD-1 Antibody Plus Chidamide and Rituximab

INTERVENTIONS:
Drug: Anti-PD-1 Antibody Plus Chidamide and Rituximab — Anti-PD-1 Antibody 200mg, ivd, D1, every 3 weeks Chidamide 30mg, po,D-1, 4, 8, 11, 15, 18, every 3 weeks Rituximab 375mg/m2, ivd, D1, every 3 weeks

SUMMARY:
To assess the efficacy and safety of Anti-PD-1 Antibody Plus Chidamide and Rituximab Regimen in the Treatment of Relapsed or Refractory DLBCL

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients: 60-75 years old.
* Relapsed or Refractory patients
* Histologically confirmed DLBCL with CD20 positive
* ECOG physical condition score: 0-1 points for patients.
* The patients must be with at least one evaluable or measurable lesion meeting LYRIC 2016 criteria.
* Patients who had received at least 2 cycles of standard first-line rituximab regimens didn't obtain remission or relapsed after remission, or who were unable or unwilling to receive chemotherapy due to illness or severe chemotherapy toxicity.
* Hematology values must be within the following limits at baseline:

  1. Absolute neutrophil count (ANC) ≥1,500 cells/μL. In case bone marrow involvement, ANC≥1,000 cells/μL.
  2. Platelets≥75,000 cells/μL. In case bone marrow involvement, platelets≥50,000 cells/μL
  3. Hemoglobin≥90 g/L.In case bone marrow involvement, hemoglobin≥70 g/L
* Biochemical values must be within the following limits at baseline:

  1. Alanine aminotransferase#ALT#≤2.5×upper limit of normal (ULN).
  2. Aspartate aminotransferase (AST) ≤2.5×ULN
  3. Total bilirubin≤1.5×ULN, unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
  4. Serum creatinine ≤2×ULN.
* LVEF ≥50%, as determined by echocardiography.
* Each subject (or their legally acceptable representative) must sigh an informed consent form (ICF) indicating that he or she understands the purpose of any procedures for the study and are willing to participate in the study.
* Thyroid stimulating hormone (TSH) or free Thyroxine (FT4) or free Triiodothyronine (FT3) were within the normal range of ±10%.
* Expected survival time ≥6 months.
* No radiotherapy, chemotherapy, targeted therapy or hematopoietic stem cell transplantation within 4 weeks before medication.

Exclusion Criteria:

* Patients with clinically symptomatic CNS metastases (e.g., cerebral edema, need for hormonal intervention, or progression of BRAIN metastases) and/or cancerous meningitis.
* A history of severe allergies or allergic reactions to drugs mentioned above.
* Patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix.
* History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome.
* Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 1000 IU/mL) andHCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 1000 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group.
* Inability to swallow, intestinal obstruction, or other factors that affect drug administration and absorption.
* Received systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc..
* Received major surgery within 28 days before treatment or radiotherapy within 90 days before treatment.
* Received live vaccination (except influenza attenuated vaccine) within 28 days before treatment.
* Patients requiring long-term systemic glucocorticoid therapy or other immunosuppressive therapy. Allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy.
* Patients suffering from uncontrollable comorbid diseases, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or bleeding disorders.
* Pregnant or lactating women.
* Patients with a history of interstitial lung disease or non-infectious pneumonia. Subjects who have previously had drug-induced or radioactive non-infectious pneumonia but asymptomatic are allowed to enroll.
* Any life-threatening disease, physical condition or organ dysfunction according to the researchers' judgment may endanger the safety of the subject or put the clinical research at excessive risk.
* Any other conditinons that the investigator considers inappropriate for participation in this study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 24 weeks
Objective remission rate | 24 weeks
Disease Control Rate | 24 weeks
Partial Remission Rate | 24 weeks

SECONDARY OUTCOMES:
Progression-free Survival | 2 years
  PFS was defined as time from study registration to first disease progression or death whichever occurred first, otherwise subject data were censored at time last known disease free
Overall Survival | 2 years
  OS was defined as time from study registration to death, and otherwise censored at time last known alive
Percentage of Participants With Adverse Events (AEs) | Up to 30 days after the last cycle of per-protocol treatment and 90 days after last dose of anti-PD-1 antibody
  Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.01

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, professor, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No